CLINICAL TRIAL: NCT06027463
Title: The Predictive Value of Clinical Data on Perioperative and Postoperative Risk Events in Patients With Head and Neck Artery Stenosis
Status: Suspended | Type: Observational
Why Stopped: paper is done, but not published.
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: liubei
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Postoperative Risk Factors for Patients With Carotid Artery Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- xi'an/Tangdu hospital
  Interventions: Procedure: Head and neck vascular recanalization

INTERVENTIONS:
Procedure: Head and neck vascular recanalization — Head and neck vascular recanalization

SUMMARY:
The Predictive Value of Clinical Data on Perioperative and Postoperative Risk Events in Patients With Head and Neck Artery Stenosis

ELIGIBILITY:
Inclusion Criteria:

* (1) All enrolled patients were diagnosed with clear head and neck artery stenosis and a risk event after head and neck revascularization;

  (2) Location of lesion: origin of internal carotid artery, bifurcation of internal and external carotid arteries;

  (3) Patients with symptomatic head and neck artery stenosis and dangerous events after head and neck blood flow reconstruction, and with a degree of stenosis ≥ 70% on non-invasive examination or stenosis ≥ 50% found on angiography;

  (4) Asymptomatic head and neck artery stenosis and risk events after head and neck revascularization, with a degree of stenosis ≥ 70% on non-invasive examination or stenosis ≥ 60% found on angiography;

  (5) Asymptomatic head and neck artery stenosis and dangerous events after head and neck blood flow reconstruction, with a non-invasive examination of stenosis degree less than 70%, but angiography or other examinations indicate that the stenosis lesion is in an unstable state;

  (6) Symptomatic head and neck artery stenosis and risk events after head and neck revascularization, non-invasive examination of head and neck artery stenosis and risk event degree after head and neck revascularization at 50% to 69%

Exclusion Criteria:

* (1) Patients with poor overall condition and intolerance to general anesthesia;

  (2) Patients with mental illness or severe mental illness;

  (3) Severe respiratory system diseases;

  (4) Pregnant and lactating women;

  (5) Participating in another clinical study;

  (6) Patients with advanced tumors or those who are expected to die within one year;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The target population of the study is adults aged 18-90 who have been diagnosed with head and neck artery stenosis and risk events after head and neck revascularization and seek medical treatment in neurosurgery departments of tertiary comprehensive hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of cerebral infarction | half a year
  Postoperative recurrence of cerebral infarction in patients

SECONDARY OUTCOMES:
Death | one year
  Patients who died after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China